CLINICAL TRIAL: NCT03388151
Title: Effect of Use of Propofol Versus Use of Midazolam as Sedative Agent in Patients With Liver Cirrhosis Presented for Lower Gastrointestinal Endoscopy, Randomised Controlled Trial
Brief Title: Propofol Versus Midazolam for Lower Gastrointestinal Endoscopy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, PhDTropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Propofol colonoscopy
Record Dates: First submitted 2017-12-23; First posted 2018-01-02 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Cirrhosis, Liver
MeSH Terms: conditions — Liver Cirrhosis | interventions — Midazolam; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midazolam (Active Comparator): Midazolam 3 mg i.v added to fentanyl 0.5 ug/kg till reaching satisfactory level of sedation
  Interventions: Drug: Midazolam
- Propofol (Active Comparator): Propofol 1 mg/kg i.v added to fentanyl 0.5 ug/kg i.v till reaching satisfactory level of sedation
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Midazolam — Midazolam 3 mg i.v added to fentanyl 0.5 ug/kg till reaching satisfactory level of sedation
  Arms: Midazolam
Drug: Propofol — Propofol 1 mg/kg i.v added to fentanyl 0.5 ug/kg i.v till reaching satisfactory level of sedation
  Arms: Propofol

SUMMARY:
propofol versus use of midazolam as sedative agent in patients with liver cirrhosis presented for lower gastrointestinal endoscopy

DETAILED DESCRIPTION:
Effect of use of propofol versus use of midazolam as sedative agent in patients with liver cirrhosis presented for lower gastrointestinal endoscopy, Randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis
* presented to colonoscopy

Exclusion Criteria:

* Encephalopathy
* Hypersensitivity
* Coagulopathy

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-04-01 (Actual); Primary Completion 2022-11-11 (Estimated); Study Completion 2022-12-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients adequately sedated | 6 months
  The number of patients adequately sedated

CONTACTS AND LOCATIONS:
Overall Officials: Sherief Abd-Elsalam, MD, Principal Investigator — Gastroenterology; Sameh Abdelkhalek Ahmed, MD, Study Director — Tanta University Anasthesia Department
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt